CLINICAL TRIAL: NCT02112578
Title: " National, Phase III, Radomized, Double-Blind, Double -Dummy, Controlled, Parallel to Evaluate Non Inferiority of Meclin® (Meclizine Chlorhydrate) Versus Dramin® (Dimenhydrinate) Soft Gel Capsules in the Control of Acute Vertigo Symphtoms From Peripheral Origin"
Brief Title: Non Inferiority of Meclin® (Meclizine Chlorhydrate) Versus Dramin® (Dimenhydrinate) in Control of Acute Vertigo Symptoms From Peripheral Origin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Apsen Farmaceutica S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APS 002/2013; BRA15APS002-2015 (Other: Apsen); U1111-1149-6768 (Other Grant/Funding Number: World Health Organization)
Record Dates: First submitted 2014-04-10; First posted 2014-04-14 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Vertigo, Peripheral
Keywords: Vertigo, Meclizine, dimenhydrinate, Peripheral Origin
MeSH Terms: conditions — Vertigo | interventions — Meclizine; Dimenhydrinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Meclizine (Experimental): Meclizine 25 mg, tablets
  Interventions: Drug: Meclizine
- Dimenhydrinate (Active Comparator): Dimenhydrinate 50 mg, soft Capsgel
  Interventions: Drug: Dimenhydrinate

INTERVENTIONS:
Drug: Meclizine — 25 mg, 3 times per day up to 30 days
  Other Names: Meclin
  Arms: Meclizine
Drug: Dimenhydrinate — 50 mg, 3 times per day up to 30 days
  Other Names: Dramin
  Arms: Dimenhydrinate

SUMMARY:
* Evaluation of the non inferiority of Meclin (meclizine) versus Dramin (Dimenhydrinate) to treat the symptoms of acute vertigo from peripheral origin after up to 4 weeks of treatment;
* Evaluation of impact on quality of life in vertigo;
* Compare the intensity of daytime sleepiness in the two treatment groups;
* Compare the efficacy of drugs in relieving each of the 10 symptoms that make up the VS;
* Compare the duration of treatment in both treatment groups;
* Compare Adehence;
* Compare the level of satisfaction from each group from the investigators and the subjects;
* Adverse events;

DETAILED DESCRIPTION:
It is a prospective interventional study arms parallel , active -controlled , non-inferiority . Participants selected for the study should be of both sexes , aged over 18 years and less than 65, which meet all the inclusion criteria and did not fit any exclusion criteria , and agree to all the purposes of the study. Participants are divided into two according to the randomization treatment groups 1:1.

The study should take no longer than 30 days to be completed with the amount of 6 visits (7±2 days): V0 radomization; V1, V2, V3 andV4(FV) are Evaluation visits and One Follow up visit 7±2 days after the Final Visit.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged over 18 years and less than 65;
* Presence of vertigo episodes of vestibular origin (peripheral ) of moderate intensity , strong or very strong according to the VS range ;
* Participants who are able to swallow tablets / capsules;
* Participants able to understand the guidance and care of this study and cooperative ;
* Participants with the requisite understanding, in accordance with Good Clinical Practice Research Document of the Americas.

Exclusion Criteria:

* Use of meclizine or dimenidrynate in the actual event or in the past 15 days;
* Use of alcohol in the past 48 hours;
* Presence of vomiting which prevent the ingestion of tablets;
* Pregnancy or breastfeeding;
* Presence of clinical condition that determines contraindication to the active substances : convulsions , suspected intracranial compressive processes , closed-angle glaucoma , prostatic adenoma with urinary disorders , liver diseases , endocrine , renal, and / or uncontrolled cardiovascular , Parkinson's disease, porphyria, know history of hipersensibility to the Actives or Excipients from the study medications;
* Malignancies History , even if no evidence of active disease for less than five years . Those without active disease for more than five years may be included;
* Uncontrolled systemic arterial hypertension ( > 140/90 mmHg );
* Decompensated diabetes mellitus (blood glucose at any time > 200 mg / dL );
* Participants with asthma or chronic obstructive pulmonary disease;
* Participants making use of antihistamines with anti-vertigo effect ( betahistine, meclizine , diphenidol ) , drugs with antagonist calcium channel action ( cinnarizine , flunarizine ) , anticholinergic drugs ( metoclopramide , dimenhydrinate , meclizine , diphenidol , scopolamine, ondansetron, granisetron ) , antiseizure drugs ( diazepam , clonazepam , carbamazepine ) and other central nervous system depressants;
* Participants with central origin vertigo or non-vestibular;
* Participants with positional benign positional paroxysmal vertigo (bppv).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Vertigo Score (VS) | up to 30 days
  Evaluation of non inferiority by measuring 10 symptoms of vertigo : distasia and instability when walking ; totter ; spinning sensation; tendency to fall; Continuous floating feeling ; floating sensation to change position ; floating sensation to bow down ; floating sensation when standing up ; floating sensation traveling on any means of transport; floating sensation with head movement ; floating sensation with eye movement. Each symptom is graduated in a semi -quantitative 5-point scale : 0 = no symptoms ; 1 = mild symptoms ; 2 = moderate symptoms ; 3 = strong symptoms ; 4 = very strong symptoms in all visits that the subject accomplishes.

SECONDARY OUTCOMES:
Quality of Life Questionnaire DHI - Dizziness Handicap Inventory, validated for the Brazilian population | up to 30 days
  Evaluation of life quality

OTHER OUTCOMES:
Stanford and Epworth Sleepiness Scale | up to 30 days
  Evaluation of somnolence (baseline measurement)
Variation of the intensity of each of the 10 symptoms | up to 30 days
  Evaluation of the variation of the intensity of each of the 10 symptoms that make up VS, along the visits
Duration of treatment (days from V0) | up to 30 days
  Evaluation of the duration of tratement from each group
Adherence rate to treatment | up to 30 days
  Evaluation of adherence rate from each group throughout the study
Visual analogue scale (VAS) for subjects and for investigators | up to 30 days
  For the subjective assessment of the participant and investigator's research on the treatment applied in 1,2,3 visits and final (VF);
Participants Percentage with any symptoms classified as moderate (score ≥2) | Since last Visit
  Evaluation of participants percentage with any symptoms classified as moderate on the VS Scale on the follow-up visit, held 7 ± 2 days after the final inspection (VF).
  through the study.
Analysis of Adverse Events | After the signature of SICF
  Evaluation of any Adverse Event ou Serious Adverse Event recorded after the signing of the Informed Consent ( IC) and until the end of the study
Clinical and Physical findings | After the signature of SICF
  Evaluation of any changes in clinical / physical assessment findings since baseline

CONTACTS AND LOCATIONS:
Overall Officials: Norton Sayeg, PhD, Principal Investigator — CCBR SP
Locations (7):
- Brazil (7):
  - Clinilive, Maringá, Paraná
  - Alergoalpha, Barueri, São Paulo
  - Pesquisare Saude S/S Ltda, Santo André, São Paulo
  - ISPEM, São José dos Campos, São Paulo
  - Irmandade da Santa Casa de Misericórdia de São Paulo, São Paulo, São Paulo
  - Clinica de Alergia MarttiAntila, Sorocaba, São Paulo
  - CCBR SP, São Paulo

IPD SHARING:
Plan to Share IPD: No